CLINICAL TRIAL: NCT06162208
Title: Examining the Effect of Action Observation Therapy Added to the Telerehabilitation-Based Standard Exercise Program on Patient-Reported and Performance-Based Outcomes in Patients Undergoing Total Knee Arthroplasty Surgery
Brief Title: Action Observation Therapy Via Telerehabilitation on Total Knee Arthroplasty Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Nihal BÜKER, Proffesor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-60116787-020-39072
Record Dates: First submitted 2023-12-01; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Knee Arthroplasty, Total; Telerehabilitation
Keywords: Telerehabilitation; Action Observation Therapy; Total Knee Arthroplasty; Patient-Reported Outcomes; Performance-Based Outcomes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home exercise group with information leaflet (No Intervention): These patients will be asked to do the exercises in the information leaflet themselves at home.
- İnformation brochure+standard exercise program group based on telerehabilitation (Active Comparator): Patients in this group will be followed up with telerehabilitation method accompanied by a physiotherapist for 30 minutes 3 times a week for 6 weeks after discharge.
  Interventions: Other: Standard exercise program based on telerehabilitation
- İnformation brochure+standard exercise program+action observation therapy group. (Active Comparator): Patients in this group will be followed up with telerehabilitation method accompanied by a physiotherapist for 30 minutes 3 times a week for 6 weeks after discharge. In addition, 15 minutes of movement observation therapy will be applied via video conferencing 3 days a week.
  Interventions: Other: Standard exercise program based on telerehabilitation

INTERVENTIONS:
Other: Standard exercise program based on telerehabilitation — Exercises included in a standard exercise program based on telerehabilitation; Week 0-3 Patellar mobilization Isometric quadriceps femoris exercise Terminal extension exercise Active assisted knee flexion Straight leg lift Active hip abduction Active assisted knee flexion in sitting SAFTE Cold pack application Week 3-6 Straight leg raises with weights Hip abduction in weighted side lying Knee flexion in the prone position Knee extension in weight-bearing sitting Sliding forward in the chair to increase the knee flexion angle Standing weighted hip abduction Standing knee flexion with weight Squat Walking Climbing stairs Action observation therapy will be practiced by watching videos of all exercises with a focus on close-up action.
  Other Names: Action observation therapy added to a standard exercise program based on telerehabilitation
  Arms: İnformation brochure+standard exercise program group based on telerehabilitation; İnformation brochure+standard exercise program+action observation therapy group.

SUMMARY:
The goal of this clinical trial is to compare patient-reported and performance-based outcomes of patients followed with a standard exercise program based on telerehabilitation and patients followed with action observation therapy program added to a standard exercise program based on telerehabilitation after total knee arthroplasty surgery.

The main questions it aims to answer are:

* [What is the effect of action observation therapy added to a telerehabilitation-based standard exercise program on patient-reported outcomes after total knee arthroplasty surgery?]
* [What is the effect of action observation therapy added to a telerehabilitation-based standardized exercise program on performance-based outcomes after total knee arthroplasty surgery?]

Participants will be divided into three groups by computer-assisted randomization method: Group 1: home exercise with information leaflet group, Group 2: information leaflet + telerehabilitation-based standard exercise program group, Group 3: information leaflet + telerehabilitation-based standard exercise program + action observation therapy group.

Patients in the second and third groups will be followed up with the telerehabilitation method accompanied by a physiotherapist for 30 minutes 3 days a week for 6 weeks after discharge. The third group will receive a standard exercise program 3 days a week and 15 minutes of action observation therapy via video conferencing.

DETAILED DESCRIPTION:
The goal of this clinical trial is to compare patient-reported and performance-based outcomes of patients followed with a standard exercise program based on telerehabilitation and patients followed with action observation therapy program added to a standard exercise program based on telerehabilitation after total knee arthroplasty surgery.

The secondary aim is to investigate the effect of a telerehabilitation-based standard exercise program added to the home program (information leaflet) on patient-reported and performance-based outcomes.

The surgical operations of all patients participating in the study will be performed by the same surgical team and a standard physiotherapy program will be applied to all patients until discharge.

Participants will be divided into three groups by computer-assisted randomization method: Group 1: home exercise with information leaflet group, Group 2: information leaflet + telerehabilitation-based standard exercise program group, Group 3: information leaflet + telerehabilitation-based standard exercise program + action observation therapy group.

Patients in the second and third groups will be followed up with the telerehabilitation method accompanied by a physiotherapist for 30 minutes 3 days a week for 6 weeks after discharge. The third group will receive a standard exercise program 3 days a week and 15 minutes of action observation therapy via video conferencing.

Telerehabilitation sessions will include information about the process and exercise training. Action observation therapy will include showing videos of the exercises in the exercise program. All patients will be evaluated before surgery and at the third, sixth, and twelfth weeks after discharge.

Evaluations

Descriptive Data: Descriptive data of the patients will be recorded using an evaluation form.

Patient Reported Assessments:

* Western Ontario McMaster University Osteoarthritis Index (WOMAC): This index questions clinically significant problems in the areas of pain, stiffness and physical function in patients with osteoarthritis of the hip and knee.
* Pain intensity: Pain intensity will be assessed with the Visual Analog Scale (VAS).
* Knee range of motion: Active and passive knee range of motion will be measured in the sitting position with a digital goniometer (HALO Medical Devices, Australia)
* Quality of Life Assessment: Knee Injury and Osteoarthritis Outcome Score - Activities of Daily Livings Scale (KOOS-ADLS) and EuroQol Group (EQ-5D) scales will be used for quality of life assessment.KOOS-ADLS is a scale used to detect symptoms and limitations in daily life tasks.The EQ-5D index scale consists of a questionnaire with five dimensions (movement, self-care, usual activities, pain/discomfort and anxiety/depression).
* Physical activity assessment: International Physical Activity Survey (IPAQ-Short Form) and smart phone pedometer application (Samsung Health®) will be used for physical activity assessment. The IPAQ-Short Form consists of 7 questions asking about various degrees of physical activity and sedentary behaviors in the past 1 week.
* Patient Satisfaction Assessments: Patient satisfaction with telerehabilitation sessions will be assessed. Technical quality (such as reliability of technology, quality of audio/video synchronization, quality of image, quality of sound), achievement of treatment goals of the session and overall satisfaction with the session will be questioned.

Performance Based Assessments:

The tests recommended by the research groups of 30 seconds of sit and stand, 40 meters fast walking and stair climbing will be used.

* Lower extremity muscle strength: Lower extremity muscle strength will be assessed by 30 seconds sit and stand test.
* Walking speed: In the 40-meter walk test, the patient is asked to walk a distance of 40 meters as fast as possible and the time in seconds is recorded.
* Locomotor performance: Locomotor performance will be assessed with the stair climbing test. The patient will be asked to ascend and descend 9 steps 16-20 centimeters long stairs as quickly but safely as possible.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer
* 40 years and older
* Undergo primary unilateral total knee arthroplasty surgery after the diagnosis of osteoarthritis
* Can understand, speak and write Turkish
* Understand verbal and written information given
* Internet access
* Able to use video conferencing program

Exclusion Criteria:

* Revision total knee arthroplasty surgery
* Previous major surgery on the extremity to be operated on
* Additional comorbid diseases such as rheumatoid arthritis, cancer
* Has any engine defect that may affect performance
* With a diagnosed psychiatric disorder
* People with alcohol or drug addiction
* Hearing or visual impairment that cannot be corrected with hearing aids or glasses
* Morbidly obese (BMI > 40 kg/m2)
* Who will not be able to participate in a six-week rehabilitation program

Exclusion Criteria for Volunteers:

* Patients who did not come to follow-up after surgery for any reason,
* Patients who want to leave the study,
* Patients who are unable to continue the study due to an additional condition will be excluded from the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain, stiffness and physical function (WOMAC) | 5 minutes
  • Western Ontario McMaster University Osteoarthritis Index (WOMAC): This index questions clinically significant problems in the areas of pain, stiffness and physical function in patients with osteoarthritis of the hip and knee.
Pain intensity | 2 minutes
  Pain intensity will be assessed with the Visual Analog Scale (VAS).
Knee range of motion | 5 minutes
  Active and passive knee range of motion will be measured in the sitting position with a digital goniometer (HALO Medical Devices, Australia).
Physical activity assessment | 5 minutes
  IPAQ-Short Form and smartphone pedometer application (Samsung Health®) will be used for physical activity assessment. The IPAQ-Short Form consists of 7 questions asking about various degrees of physical activity and sedentary behaviors in the past 1 week.
Lower extremity muscle strength | 30 seconds
  Lower extremity muscle strength will be assessed by 30 seconds sit and stand test.
Walking speed | Average 5 minutes
  In the 40-meter walk test, the patient is asked to walk a distance of 40 meters as fast as possible and the time in seconds is recorded.
Locomotor performance | Average 5 minutes
  Locomotor performance will be assessed with the stair climbing test. The patient will be asked to ascend and descend 9 steps 16-20 centimeters long stairs as quickly but safely as possible.

SECONDARY OUTCOMES:
Quality of Life Assessment | 10 minutes
  KOOS-ADLS and EQ-5D scales will be used for quality of life assessment.KOOS-ADLS is a scale used to detect symptoms and limitations in daily life tasks.The EQ-5D index scale consists of a questionnaire with five dimensions (movement, self-care, usual activities, pain/discomfort and anxiety/depression).
Patient satisfaction assessment | 2 minutes
  Patient satisfaction with telerehabilitation sessions will be assessed. Technical quality (such as reliability of technology, quality of audio/video synchronization, quality of image, quality of sound), achievement of treatment goals of the session and overall satisfaction with the session will be questioned.

CONTACTS AND LOCATIONS:
Overall Officials: Sinem Yenil, Msc, PT, Principal Investigator — Pamukkale University; Harun Reşit Güngör, Prof., Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Villafane JH, Isgro M, Borsatti M, Berjano P, Pirali C, Negrini S. Effects of action observation treatment in recovery after total knee replacement: a prospective clinical trial. Clin Rehabil. 2017 Mar;31(3):361-368. doi: 10.1177/0269215516642605. Epub 2016 Jul 10. PMID 27068367
- [Background] Windsor EN, Sharma AK, Gkiatas I, Elbuluk AM, Sculco PK, Vigdorchik JM. An Overview of Telehealth in Total Joint Arthroplasty. HSS J. 2021 Feb;17(1):51-58. doi: 10.1177/1556331620972629. Epub 2021 Feb 21. PMID 33967642
- [Background] McKeon JF, Alvarez PM, Vajapey AS, Sarac N, Spitzer AI, Vajapey SP. Expanding Role of Technology in Rehabilitation After Lower-Extremity Joint Replacement: A Systematic Review. JBJS Rev. 2021 Sep 13;9(9). doi: 10.2106/JBJS.RVW.21.00016. PMID 34516463